CLINICAL TRIAL: NCT02018003
Title: The Effect of Postoperative Therapy on the Quality of Life of Patients With Early Stage Cervical Cancer
Brief Title: The Effect of Postoperative Therapy on the Quality of Life of Patients With Early Cervical Cancer Research
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Yunong Gao, the head of department of gynecological oncology, Peking University
Other Study IDs: PUCRP201309
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-11

CONDITIONS: Uterine Cervical Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to assess the women's quality of life, who accepted chemotherapy,radiotherapy, concurrent radiochemotherapy or who didn't accept therapy, after operation.

DETAILED DESCRIPTION:
The study projects to follow up 180-200 early stage cervical cancer patients after operation and assess the women's quality of life by the scales: ECOG, Functional Assessment of Cancer Therapy, EuroQol-5 Dimensions, and Kupperman index.

ELIGIBILITY:
Inclusion Criteria:

* ≮ 18 years, cervical cancer verified by pathology，

  * IIA stage, accepted the operation ( Piver III and pelvic lymph node dissection) as initial therapy， obtained the patient's agreement

Exclusion Criteria:

* the patient had accepted chemotherapy or radiotherapy before operation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The women with early stage cervical cancer, who underwent operation in Peking University School of Oncology.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life for the women with early stage cervical cancer who underwent operation | up to 12 months after operation

CONTACTS AND LOCATIONS:
Overall Officials: Gao Yunong, Study Director — Peking University